CLINICAL TRIAL: NCT06398899
Title: Sugammadex Compared With Neostigmine/Glycopyrrolate in Impact of Postoperative Urinary Retention for ENT Surgery Patients With High-risk of Dysuria
Brief Title: Sugammadex v.s. Neostigmine/Glycopyrrolate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202307081MINA
Record Dates: First submitted 2024-03-05; First posted 2024-05-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Surgery; Chronic Sinusitis; Chronic Otitis Media; Laryngeal Disease
Keywords: Sugammadex; anticholinergic drug; postoperative urinary retention; ENT surgery; neostigmine
MeSH Terms: conditions — Laryngeal Diseases | interventions — Sugammadex; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Sugammadex or Neostigmine/Glycopyrrolate
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S (Experimental): Sugammadex as reversal agent
  Interventions: Drug: Group S: sugammadex injection
- Group N (Active Comparator): neostigmine and glycopyrrolate as reversal agent
  Interventions: Drug: Group N: neostigmine/glycopyrrolate

INTERVENTIONS:
Drug: Group S: sugammadex injection — Reversal agent: sugammadex
  Other Names: Bridion
  Arms: Group S
Drug: Group N: neostigmine/glycopyrrolate — Reversal agent: glycopyrrolate and neostigmine
  Other Names: vagostin injection/glycopyrodyn
  Arms: Group N

SUMMARY:
The aim of study is to clarify the role of sugammadex in ENT surgery patients with a prior history of postoperative urinary retention, benign prostatic hypertrophy, or a history of prostate cancer, to prevent postoperative urinary retention. The main question it aims to answer are:

* Anticholinergic agent interferes the postoperative urination
* Sugammadex does not interfere postoperative urination Sugammadex can be recommended for these patients with high risk in postoperative urinary retention in the future.

DETAILED DESCRIPTION:
Investigators will evaluate the benefit of sugammadex in reducing postoperative urinary retention for these head and neck surgery patients with high-risk for dysuria. The definition of high-risk of dysuria is patient with a prior history of urinary retention, benign prostatic hypertrophy, or a history of prostate cancer.

Patients scheduled to undergo ENT surgery within Three hours of expected surgical time are enrolled. These patients are associated with high-risk of postoperative urinary retention, including prior history of postoperative urinary retention, benign prostatic hypertrophy, or a history of prostate cancer. They are randomly divided these patients into sugammadex group (Group S) and neostigmine/glycopyrrolate group (Group N), sugammadex or neostigmine/glycopyrrolate are used during recovery period of anesthesia, to compare the incidences of postoperative urinary retention, nausea/vomiting, bradycardia, hypotension, and dry mouth in these patients after ENT surgery. Sugammadex can be recommended for these high-risk patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* ENT surgery patients whose surgery is expected to take less than three hours and no planned Foley catheter
* high risk of postoperative urinary retention, including

  * prior history of postoperative urinary retention
  * benign prostatic hypertrophy
  * history of prostate cancer

Exclusion Criteria:

* refusal or inability to provide informed consent
* age younger than 18 years
* American Society of Anesthesiologists class more than III
* pregnancy
* impaired renal function (creatinine clearance < 30 mL/min)
* allergy to a study drug

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
postoperative urinary retention | up to 48 hours
  Postoperative urinary retention is defined as patient discomfort or a palpable bladder, with a bladder volume of ≥400 mL confirmed by bladder scan or catheterization, requiring intervention.

SECONDARY OUTCOMES:
postoperative nausea and vomiting | 48 hours
  postoperative nausea and vomiting
bradycardia | 24 hours
  Bradycardia was defined as a heart rate of less than 50 beats per minute.
thirsty intensity | 24 hour
  thirsty intensity during postanesthesia care unit
length of hospital stay | during admission (assessed up to 7 days)
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: PEILIN LN, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan